CLINICAL TRIAL: NCT01894282
Title: Mind Body Intervention for Chronic Lower Back Pain: A Pilot Study
Brief Title: Mind Body Intervention for Chronic Lower Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Dougherty, DC, Chiropractor, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBI001
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Lower Back Pain
Keywords: Chronic Lower Back Pain; Manual Therapy; Cognitive Behavioral Therapy
MeSH Terms: interventions — Musculoskeletal Manipulations; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy (Active Comparator): Spinal Manipulative therapy (SMT) for the purpose of this study we will allow the use of other types of MT, including non-thrust spinal mobilization and flexion-distraction technique.
  Interventions: Procedure: Manual Therapy
- Mind Body Intervention (MBI) (Experimental): Mind Body Intervention will consist of a combination of the previously described "manual therapy" and Cognitive Behavioral Therapy for pain (CBT-p). Cognitive Behavioral Therapy for pain management has three basic components. The treatment rationale, coping skills training and application and maintenance of learned coping skills.
  Interventions: Procedure: Manual Therapy; Procedure: Mind Body Intervention

INTERVENTIONS:
Procedure: Manual Therapy — Manual Therapy Arm
  Other Names: Spinal Manipulative Therapy; Spinal Mobilization; Flexion Distraction Therapy
Procedure: Mind Body Intervention — Combination of manual therapy and cognitive behavioral therapy for pain.
  Other Names: Manual Therapy; Cognitive Behavioral Therapy for Pain
  Arms: Mind Body Intervention (MBI)

SUMMARY:
This pilot study will evaluate the feasibility of having a non-behavioral health provider deliver a combination of manual therapy (MT) and cognitive behavioral therapy for pain (CBT-p). In addition, we will evaluate differences in outcomes in patients undergoing the combined intervention of CBT-p and MT and those undergoing MT alone.

DETAILED DESCRIPTION:
Given that this is a pilot study we will use simple descriptive statistics for patient characteristics, including age, sex, BMI and baseline scores on outcome measures. In addition we will assess the inter-rater reliability of the scoring of the delivery of the CBT-p by the two trained practitioners utilizing kappa statistics. We will perform data analyses using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 69 years of age with CLBP who are
* "high risk" for poor prognosis based on SBST
* currently undergoing chiropractic care.

Exclusion Criteria:

* Contraindications to either MT or CBT-p.
* Patients who are currently undergoing CBT-p
* who have been treated for substance abuse in the past year.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline and 6 weeks post baseline (immediately post intervention)
  The VAS is a patient completed analogue measure that evaluates pain intensity on a 100 mm long horizontal line, which is anchored at each end with a statement representing the extremes of the dimension being measured. In this case the left hand side reads, "no pain" and the right hand side reads "worst pain possible". The VAS scale utilized will assess pain at the current time. The VAS has been established as a reliable, valid and generalizable measure that can be administered in a wide range of clinical and experimental settings.

SECONDARY OUTCOMES:
PROMIS Global Health Scale (GHS) | Baseline and 6 weeks post baseline (immediately post intervention)
  Health outcomes assessment has advanced to a point where generic health-related quality of life (HRQL) measures are often used to examine the health status of populations and the effects of medical interventions. Generic HRQL profile measures, such as the SF-36 Health Survey, provide multiple health domains scores (e.g., physical function, mental health, pain, vitality, etc.), but not an overall index score. Patient reported outcome measurement information system has developed a quality of life tool that provides an overall index score for quality of life. The main advantage of the PROMIS measures over other static health status measures is that the PROMIS domain item banks and scores allow flexibility in administration using either targeted short forms or computerized adaptive testing. This form has recently been validated in comparison to the EuroQual.

OTHER OUTCOMES:
Patient Satisfaction Questionnaire | Baseline and post intervention
  Cherkin et al, in the evaluation of a physician education program developed a patient satisfaction questionnaire which was found to be reliable and valid. The questionnaire utilized in this study will incorporate these same questions. Additional questions to be included focus on the burden of the data collection activities, and suggestions for subject recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dougherty, DC, Principal Investigator — Canandaigua VA Medical Center
Locations (1):
- Rochester Outpatient Clinic, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided